CLINICAL TRIAL: NCT04336345
Title: Outcomes of Patients With COVID-19 in the Intensive Care Unit: A National Observational Study (Mexico COVID-19 ICU Study)
Brief Title: Outcomes of Patients With COVID-19 in the Intensive Care Unit
Acronym: MexCOVID-19
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Silvio A. Ñamendys-Silva, Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Other Study IDs: 3336
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Coronavirus Infections; COVID-19; Viral Pneumonia Human Coronavirus
Keywords: Intensive care unit; Critical care; Outcomes; Epidemiology
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the clinical characteristics and outcomes of critically ill patients with COVID-19 admitted to the intensive care unit.

A Multicenter Observational Study.

DETAILED DESCRIPTION:
As of 23 March 2020, a cumulative total of 332,930 confirmed cases of coronavirus disease 2019 (COVID-19) were reported in 189 countries and territories worldwide. As of this time, there had been 367 total confirmed cases of COVID-19, including four deaths in Mexico. The clinical manifestations of patients with COVID-19 are wide, asymptomatic infection, mild upper respiratory tract illness, and approximately 5% of critically ill patients with COVID-19 have presented rapidly progressive respiratory failure, development of acute respiratory distress syndrome (ARDS), and intensive care unit (ICU) admission. On March 24, 2020, the Secretary of Health of Mexico, formally declared the beginning of phase 2. It has been estimated that many confirmed cases of COVID-19 would occur, thus would result in a significant increase of hospital and ICU admissions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed case: Critically ill patient who meets the operational definition of a suspected case and who has a confirmed diagnosis by the National Network of Public Health Laboratories recognized by the Institute of Epidemiological Diagnosis and Reference (Indre) (Mexico).

Exclusion Criteria:

* If a negative for SARS-CoV-2 result is obtained from a critically ill patient with a high index of suspicion for COVID-19 virus infection.
* Patients who had participated in another observational study in the last 30 days prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients aged over 18 years with a positive for SARS-CoV-2 result required admission to an intensive care unit or critical care in other areas of the hospital (critical care surge capacity).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 30 days
  Mortality 30 days following hospital admission

SECONDARY OUTCOMES:
Length of stay in the intensive care unit | Through study completion, an average of 30 days
  The number of calendar days from the day of admission (counted as 1 day) to day of intensive care unit discharge

CONTACTS AND LOCATIONS:
Overall Officials: Silvio A. Ñamendys-Silva, MD, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Guillermo Dominguez-Cherit, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Eduardo Rivero-Sigarroa, MD, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (2):
- Mexico (2):
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City
  - All centres from Mexico willing to contribute are Welcome., México

IPD SHARING:
Plan to Share IPD: Undecided
All IPD that underlie could results in a publication.

REFERENCES:
- [Result] Namendys-Silva SA, Alvarado-Avila PE, Dominguez-Cherit G, Rivero-Sigarroa E, Sanchez-Hurtado LA, Gutierrez-Villasenor A, Romero-Gonzalez JP, Rodriguez-Bautista H, Garcia-Briones A, Garnica-Camacho CE, Cruz-Ruiz NG, Gonzalez-Herrera MO, Garcia-Guillen FJ, Guerrero-Gutierrez MA, Salmeron-Gonzalez JD, Romero-Gutierrez L, Canto-Castro JL, Cervantes VH; Mexico COVID-19 Critical Care Collaborative Group. Outcomes of patients with COVID-19 in the intensive care unit in Mexico: A multicenter observational study. Heart Lung. 2021 Jan-Feb;50(1):28-32. doi: 10.1016/j.hrtlng.2020.10.013. Epub 2020 Oct 21. PMID 33138974